CLINICAL TRIAL: NCT04312906
Title: A Baseline Study in Support of Clinical Evaluation of an Oral Shigella Vaccine Development in Africa
Acronym: ShigOraVax
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: European Vaccine Initiative (Other); Groupe de Recherche Action en Sante (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: ShigOraVax Epi
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diarrhea; Diarrhea Infectious
Keywords: diarrhea; Shigella; Vaccine
MeSH Terms: conditions — Diarrhea; Dysentery; Dysentery, Bacillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool- Isolates will be grown on horse blood agar and Shigella Salmonella agar plates overnight at 37°C to detect potential contamination. Only pure ETEC and Shigella cultures will be used for DNA extraction. For Illumina whole genome sequencing, we will use the Genomic DNA kit (Promega) for DNA extraction according to the manufacturer's instructions. For Single-Molecule Real Time (SMRT) sequencing (Pacific Bioscience) which requires long intact strands of DNA, we will use the phenol-chloroform extraction method described by Mentzer and others (2014). The DNA will be stored in E buffer and sequenced at the Wellcome Trust Sanger Institute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
This study aims to address the paucity of accurate incidence data of diarrheal diseases associated with Shigella in Zambia and Burkina Faso. Given the limited feasibility of the current complex diagnostic methods used to detect Shigella in endemic and developing countries due to the costs, the none availability of reagents and a requirement of expensive and complex machinery, we suggest to use a rapide, easy-to-use, cost-effective, and robust Polymerase Chain Reaction (PCR) based rapid tool, the Loop-mediated isothermal amplification (LAMP) based diagnostic assay (ES-RLDT). This baseline study will enable us to generate an accurate estimate of Shigella incidence so as to inform future trials' designs of an oral vaccine development (ShigOraVax) in Burkina Faso and Zambia.

This project is part of the EDCTP2 programme supported by the European Union under grant agreement "No RIA2018V-2308

DETAILED DESCRIPTION:
This is an observational, cohort study to determine the incidence of Shigella in children under 5 years in Zambia and Burkina Faso.

We will first identify the population at risk i.e children that will form the cohort of children to be followed up in the study. In Zambia, this will be done through a household census that will be conducted to identify children under 5 years in the catchment areas served by the selected health facility. In Burkina Faso, the study will be conducted in the Ouagadougou Health and Demographic Surveillance System (OHDSS) catchment area. Children under five years old will be randomly selected from the OHDSS database. The heads of households or guardians of the randomly selected children will be approached for the informed consenting process to enrol into the cohort study.

We will then follow up these children using active and passive surveillance systems follow for the duration of the study. During passive follow-up, a surveillance system will be set up at the selected health facilities serving the catchment populations. Parents/guardians of enrolled children will be asked to take their child to designated health facilities once they develop an episode of diarrhoea. At presentation, a clinical evaluation will be performed on the child and the data recorded. A stool sample/rectal swab will then be collected. Once a stool sample is tested positive for Shigella, the participant will be actively followed up and monitored on days 3, 5, 7 and 9 to inquire about the disease outcome and to collect blood and stool samples.

Active follow-ups will include a combined home and clinic visits. The parents or guardians of participants enrolled in the study will be contacted through phone calls and/or home visits by trained study staff every month to collect information on the child health status. They will enquire on whether the child had an episode of diarrhoea and fever in the preceding four weeks, the use of healthcare services for the diarrhoea episode and any treatment received for the diarrhoea and fever. If an episode of diarrhoea is detected during any of the active visits, the parents/guardians will be encouraged to take the child to the clinic for appropriate management. The child will then go through the passive surveillance procedures.

MSD cases will be defined as a three or more loose stools or at least one bloody/mucoid stool within a 24 hour period (WHO, 2005). A diarrhoea episode will be defined as new if the diarrhea definition is met after seven days free of diarrhoea or dysentery. A Shigella case will be defined as any loose stool with LAMP confirmed Shigella.

In Ndola, the burden of shigella disease will be determined in under five children presenting with moderate to severe diarrhea and admitted to Arthur Davison children's hospital in Ndola.

ELIGIBILITY:
Inclusion Criteria:

* Children who are under five years, are resident in the catchment areas of participating health facilities and whose parents or guardians have no anticipated plan to leave the area for the next 12 months;
* Willing to submit child biological samples for testing and/or storage;
* Parent or guardian providing written informed consenting to the study.

Exclusion Criteria:

* Any child born after the Census has taken place(Zambia) or whose household was not randomly selected from the database (Burkina Faso)
* Current participation in a research with the use of any drug or vaccine.
* Parent or guardian unwilling to provide consent
* Any confirmed or suspected immunosuppressive or immuniodeficiency condition based on medical history and physical examination (No testing will be done for HIV)
* A family history of congenital or hereditary immunodeficiency
* Major congenital defects
* Immunosuppresive therapy within 3 months prior to recruitment

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 5 years of age living in the study catchment areas
Sampling Method: Non-Probability Sample
Enrollment: 1334 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Shigella diarrheal disease in children under fives in Zambia and Burkina Faso | 1 year
  number of children testing Shigella positive during course of study

SECONDARY OUTCOMES:
Attributable fraction for Shigella among all-cause MSD in children under 5 years | 1 year
  the number of children presenting with MSD with confirmed Shigella
Incidence of ETEC diarrheal disease in children under fives in Zambia and Burkina Faso | 1 year
  the number of children presenting with MSD with confirmed ETEC
Antimicrobial susceptibility/resistance of isolates to common antibiotics | 1 year
  Proportion of shigella isolates resistant to common antibiotics
Predictive accuracy of the modified diarrhoea severity scoring tool among children presenting with MSD | 1 year
  Proportion of MSD cases confirmed by the modified severity score

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Hourard, Study Director — European Vaccine Initiative
Locations (3):
- Schiphra Hospital, Ouagadougou, Burkina Faso
- Zambia (2):
  - Arthur Davidson Childrens Hospital, Ndola, Copperbelt
  - Chainda South Health Facility, Lusaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kotloff KL, Winickoff JP, Ivanoff B, Clemens JD, Swerdlow DL, Sansonetti PJ, Adak GK, Levine MM. Global burden of Shigella infections: implications for vaccine development and implementation of control strategies. Bull World Health Organ. 1999;77(8):651-66. PMID 10516787
- [Background] Platts-Mills JA, Liu J, Rogawski ET, Kabir F, Lertsethtakarn P, Siguas M, Khan SS, Praharaj I, Murei A, Nshama R, Mujaga B, Havt A, Maciel IA, McMurry TL, Operario DJ, Taniuchi M, Gratz J, Stroup SE, Roberts JH, Kalam A, Aziz F, Qureshi S, Islam MO, Sakpaisal P, Silapong S, Yori PP, Rajendiran R, Benny B, McGrath M, McCormick BJJ, Seidman JC, Lang D, Gottlieb M, Guerrant RL, Lima AAM, Leite JP, Samie A, Bessong PO, Page N, Bodhidatta L, Mason C, Shrestha S, Kiwelu I, Mduma ER, Iqbal NT, Bhutta ZA, Ahmed T, Haque R, Kang G, Kosek MN, Houpt ER; MAL-ED Network Investigators. Use of quantitative molecular diagnostic methods to assess the aetiology, burden, and clinical characteristics of diarrhoea in children in low-resource settings: a reanalysis of the MAL-ED cohort study. Lancet Glob Health. 2018 Dec;6(12):e1309-e1318. doi: 10.1016/S2214-109X(18)30349-8. Epub 2018 Oct 1. PMID 30287127
- [Background] GBD Diarrhoeal Diseases Collaborators. Estimates of global, regional, and national morbidity, mortality, and aetiologies of diarrhoeal diseases: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Infect Dis. 2017 Sep;17(9):909-948. doi: 10.1016/S1473-3099(17)30276-1. Epub 2017 Jun 1. PMID 28579426
- [Background] Song T, Toma C, Nakasone N, Iwanaga M. Sensitive and rapid detection of Shigella and enteroinvasive Escherichia coli by a loop-mediated isothermal amplification method. FEMS Microbiol Lett. 2005 Feb 1;243(1):259-63. doi: 10.1016/j.femsle.2004.12.014. PMID 15668027
- See also: Information about the project — https://www.shigoravax.org
- See also: Information about the call — https://www.edctp.org/vaccines-for-diarrhoeal-diseases-or-lower-respiratory-tract-infections-2018/